CLINICAL TRIAL: NCT03814096
Title: Point-Of-Care Testing for Congenital Syphilis in Mothers and Newborns: A Proof of Concept Study
Brief Title: Point-Of-Care Testing for Congenital Syphilis in Mothers and Newborns
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not secured
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Principal Investigator, Despina Contopoulos-Ioannidis, Clinical Associate Professor, Department of Pediatrics, Division of Infectious Diseases, Stanford University School of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49086
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Maternal Syphilis During Pregnancy - Baby Not Yet Delivered; Congenital Syphilis
Keywords: Syphilis, prenatal screening, SHC, point-of-care test
MeSH Terms: conditions — Syphilis, Congenital; Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Syphilis POC-prenatal screening (Experimental): Syphilis prenatal screening late in gestation at 24-28 weeks (at the time of the routine prenatal care clinic visit for the routine Glucose Tolerance Test [GTT]) using the Syphilis Health Check POC-test (Diagnostics Direct LLC, NJ)
  Interventions: Diagnostic Test: Syphilis Health Check POC-test (Diagnostics Direct LLC, NJ)

INTERVENTIONS:
Diagnostic Test: Syphilis Health Check POC-test (Diagnostics Direct LLC, NJ) — Syphilis Health Check (SHC) POC-test is a treponemal POC-test based on 3d generation enzyme immunoassay (EIA) method detecting both Immunoglobulin G (IgG) and Immunoglobulin M (IgM) antibodies.

SUMMARY:
A dramatic rise in syphilis has been recently reported in the US between 2000-2017, which was followed also by a dramatic rise in congenital syphilis (CS). In 2017 there were 918 CS cases reported in the United States, including 64 syphilitic stillbirths. In 2017, California (CA) had one of the highest syphilis rates among women and this was accompanied by a dramatic increase in CS cases. Approximately 40% of CS cases in the United States occurred from maternal infections acquired late in gestation, missed by current-early gestation only-prenatal screening. More frequent prenatal screening late in gestation is urgently needed. However, cost considerations and operational logistic limitations preclude implementation even in high risk regions. There is an urgent need for widespread implementation of more frequent prenatal screening using alternative cost-saving screening approaches. The Syphilis-Health-Check (SHC) point-of-care (POC) test is a well validated POC-test that is already commercially available in the US, is approved by the Federal Drug Administration (FDA) and Clinical Laboratory Improvement Amendments (CLIA)-waived. POC prenatal syphilis screening late in gestation using a well validated POC-test (in addition to the standard early gestation-screening with laboratory-based tests) could provide a cost-saving complementary alternative that could benefit patients, mitigate the higher cost associated with more frequent testing, overcome operational limitations and contribute to the elimination of CS. Moreover, POC-neonatal and placental screening could provide an additional complementary safeguard approach to decrease missed/delayed CS diagnoses.

DETAILED DESCRIPTION:
Given the dramatic rise in syphilis that has been recently reported in the United States in the recent years (between 2000-2017) there is an urgent need for widespread implementation of more frequent prenatal syphilis screening using alternative cost-saving screening approaches. The Syphilis-Health-Check (SHC) point-of-care (POC) test is a well validated POC-test that is already commercially available in the United States, is approved by the Federal Drug Administration (FDA) and Clinical Laboratory Improvement Amendments (CLIA)-waived. Hypotheses: a) Point-Of-Care (POC) prenatal syphilis screening late in gestation using a well validated POC-test (in addition to the standard early gestation-screening with lab-based tests) could provide a cost-saving complementary alternative that could benefit patients, mitigate the higher cost associated with the need for more frequent syphilis screening, overcome operational limitations and contribute to the elimination of CS. b) POC-neonatal screening can provide additional complementary safeguard approach to decrease missed/delayed CS diagnoses. POC-neonatal syphilis screening can be used as a rapid screening tool to capture/probe all neonatal cases who would need immediate medical attention and further investigation and workup to rule out (or rule-in accordingly) suspected/probable CS.

Specific Aim 1: Validate the diagnostic accuracy of SHC-POC-test in late gestation (24-28 weeks): a) against standard laboratory based syphilis treponemal tests (TT)/and non-treponemal tests (NTT) in prenatal-care clinic settings and b) also against clinical diagnoses of maternal syphilis requiring treatment during gestation (co-primary endpoint). Specific aim 2: Test the feasibility of POC-prenatal screening (secondary endpoint) and efficacy of POC-prenatal screening to decrease the incidence of CS in a high risk region, through prompt diagnosis (and treatment accordingly) of maternal syphilis cases that need immediate treatment (to prevent mother-to -child transmission) (co-primary endpoint). Specific Aim 3: Evaluate the feasibility of POC-neonatal screening and POC-placental screening and the concordance of the results between late gestation maternal, neonatal and placental POC-test results. (Proof of concept; secondary endpoints).

Study design: (a) Prospective cohort study in the Santa Clara Valley Medical Center (SCVMC), San Jose, CA over a 3 yr study period with enrollment of pregnant women at 24-28 weeks (wks) gestational age (GA), presenting for their routine clinic visit at 24-28 wks for their glucose tolerance test (GTT). SCVMC recently introduced as a new standard of care rescreening for syphilis of all pregnant women at 24-28 wks with TT/NTTs, bundled to the venipuncture for the Glucose Tolerance Test (GTT). During this clinic visit, the syphilis POC-testing will be done via a fingerstick in clinic, while the standard lab-based syphilis screening will be done via venipuncture in the lab (as part of the new standard of care). (b) Proof-of-concept prospective cohort substudy to test the feasibility of neonatal POC-testing (whole-blood collected via heel stick, bundled with the routine newborn screening for inborn errors of metabolism at 24-48 hours of life) and placental-POC-testing.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult pregnant women between 24-28 weeks GA seen at Obstetrics/Gynecology (OB/GYN) prenatal-care clinics in Santa Clara Valley Medical Center San Jose CA, at the time of their routine clinic visit at 24-28 weeks GA for their routine glucose-tolerance-test (GTT) prenatal screening.

Exclusion Criteria:

* Non-adult pregnant patients <18 years of age and pregnant women not between 24-28 weeks gestational age at the time of the clinic visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2022-10-29 (Estimated); Study Completion 2023-10-29 (Estimated)

PRIMARY OUTCOMES:
Count of pregnant women with concordant test results between the SHC-POC test and the TT/NTT test at 24-28 weeks gestational age, as a measure of validation of the diagnostic accuracy of the SHC-POC-test | Between 24-28 weeks gestational age of study participants
  Diagnostic accuracy of SHC-POC test against standard laboratory diagnostic tests for syphilis (TT/NTT) in late gestation (24-28 weeks)
Count of pregnant women with concordant test results between the SHC-POC test and maternal syphilis diagnosis at 24-28 weeks gestational age requiring treatment during gestation, as a measure of validation of the diagnostic accuracy of the SHC-POC test | Between 24-28 weeks gestational age of study participants
  Diagnostic accuracy of SHC-POC test against maternal syphilis diagnosis late in gestation requiring treatment during gestation (24-28 weeks)
Incidence of Congenital Syphilis (N of congenital Syphilis cases/ N of total births), as a measure of efficacy of POC-prenatal syphilis screening at 24-28 weeks gestational age | At birth and up to 3 months of age of offsprings of study participants
  The efficacy of SHC-POC prenatal screening in decreasing the incidence of Congenital Syphilis will be calculated. Comparison will be made between the incidence rate of Congenital Syphilis cases before the SHC-POC-prenatal screening (among all births in Santa Clara Valley Medical Center, San Jose, CA in the year before the SHC-POC-prenatal screening) and 3 years after the implementation of the SHC POC-prenatal screening (among all births from the screened participating pregnant women)

SECONDARY OUTCOMES:
Count of concordant SHC-POC-test results between maternal, placental and neonatal SHC-POC-testing. | At 24-28 weeks gestational age of study participants (for maternal POC-test results); During Delivery (for placental POC-test results) and at birth and up to 3 months of age of offsprings of study participants (for neonatal POC-test results)
  As a proof of concept, testing with the SHC-POC test also the placenta (at the time of delivery) and the offsprings of a minimum 20 consenting pregnant women will be done. The counts of SHC-POC test results that were concordant in the mothers, placentas and newborns will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Despina G. Contopoulos-Ioannidis, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center; Department of Obstetrics & Gynecology and Pediatrics, San Jose, California
  - Stanford University School of Medicine, Department of Pediatrics, Division of Infectious Diseases, Stanford, California

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol and the study analysis plan. The informed consent forms and the database with the completely de-identified patient data (without any Personal Health Information (PHI)) will become available upon request from the study Principal Investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available within 2 years from the completion of the study and will stay available.
Access Criteria: The informed consent forms and the database with the completely de-identified patient data (without any Personal Health Information (PHI)) will become available upon request from the study Principal Investigator.